## CONSENT FORM FOR PARTICIPANTS IN RESEARCH PROJECTS





| patterns of people living with psoriasis in the UK. | | | |
|---|---|---|---|
| Ethical review reference number: LRS/DP-21/22-29257 Version number: 30/0 | | | 5/2022 |
| | | | Tick or initial |
| 1. | I confirm that I have read and understood the information sheet project. I have had the opportunity to consider the information at which have been answered to my satisfaction. | | |
| 2. I consent voluntarily to be a participant in this project and understand that I can refuse to take part and can withdraw from the project at any time, without having to give a reason, up until May 1 2023. | | | |
| | 3. I consent to the processing of my personal information for the purposes explained to me in the Information Sheet. I understand that such information will be handled under the terms of UK data protection law, including the UK General Data Protection Regulation (UK GDPR) and the Data Protection Act 2018. | | |
| 4. | I understand that my information may be subject to review by re from the College for monitoring and audit purposes. | sponsible individuals | |
| 5. | I understand that confidentiality and anonymity will be maintaine possible to identify me in any research outputs | d, and it will not be | |
| 6. | I agree that the <b>researcher/research</b> team may use my data for understand that any such use of identifiable data would be revie a research ethics committee. (In such cases, as with this project identifiable in any report). | wed and approved by | |
| 7. | I understand that I must not take part if I fall under the exclusion detailed in the information sheet. | criteria as | |
| 8. | I understand that the information I have submitted will be publish | ned as a report | |
| 9. | I wish to receive a copy of the final report. | | |
| 10 | . I agree to be re-contacted in the future by King's College Londo regarding this project. | n researchers | |
| 11. I agree that the researcher may retain my contact details so that I may be contacted in the future by King's College London researchers who would like to invite me to participate in future studies of a similar nature. | | | |

| Name of Participant | Date | Signature |
|---------------------|----------|-----------|
| Name of Researcher | <br>Date | |